CLINICAL TRIAL: NCT04595890
Title: Knee Injections for the Clinical Management of Knee OsteoArthritis
Acronym: KICK-OA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Discontinued funding
Sponsor: University of Delaware (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1893057
Record Dates: First submitted 2020-10-08; First posted 2020-10-22 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Knee Osteoarthritis
Keywords: Physical Activity; MRI; Autologous Nucleated Cells
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intervention Group (Experimental): Injection of Bone Marrow Concentrate (BMC)
  Interventions: Device: Arthrex Angel System used to prepare injection of Bone Marrow Concentrate (BMC)
- Control Group (Placebo Comparator): Injection of saline
  Interventions: Other: Saline injection

INTERVENTIONS:
Device: Arthrex Angel System used to prepare injection of Bone Marrow Concentrate (BMC) — Participants will have bone marrow aspirated from their iliac crest, then processed using the Arthrex Angel System to produce autologous bone marrow concentrate (BMC). Then, BMC will be injected into the participant's knee with knee osteoarthritis (OA).
  Arms: Intervention Group
Other: Saline injection — Participants will have bone marrow aspirated from their iliac crest to maintain masking. Then, saline will be injected into the participant's knee with knee osteoarthritis (OA).
  Arms: Control Group

SUMMARY:
Knee osteoarthritis (OA) is an incurable disease that involves breakdown of the knee joint. This breakdown is often accompanied by knee pain and stiffness, which can limit a person's daily physical activity. Fortunately, there are treatments that may stop or slow the progression of knee OA. Bone marrow aspirate can be extracted and processed into autologous, nucleated cells, then injected back into the knee affected by OA. These cells provide important nutrients that can improve the health of the knee joint and alleviate the symptoms of knee OA.

Therefore, the investigators are interested in determining whether an injection of autologous, nucleated cells can improve physical activity, pain and function in people who are diagnosed with knee OA.

The investigators will recruit a total of 100 subjects for this study and examine changes in physical activity using a research-grade Actigraph Monitor.

ELIGIBILITY:
Inclusion Criteria:

* Adults 40-79 years of age
* Doctor-diagnosed knee OA

Exclusion Criteria:

Related to knee OA diagnosis:

* Seeking treatment for end-stage knee OA (Kellgren-Lawrence Grade 4 on X-ray)
* Seeking advanced treatment options for knee OA (e.g., knee replacement) within 6 months
* Seeking treatment for bilateral symptomatic knee OA

Related to current health status or medical history:

* Findings on clinical examination that preclude safe participation in the study, including (but not limited to):

  * 3+ effusion of the target knee
  * Significant varus or valgus alignment deformity
* Non-ambulatory (e.g., use a manual or power wheelchair)
* Diagnosis of rheumatoid arthritis, inflammatory arthritis, or gout
* Uncontrolled diabetes (e.g., glycosylated hemoglobin level >7.0)
* Known contraindications to MRI, including: heart pacemaker, artificial heart valves, metal implants such as metal ear implants, bullet pieces, chemotherapy or insulin pumps, metal clips or rings
* Body mass index > 40 kg/m 2
* Increased risk for postsurgical bleeding (e.g., bleeding disorder or taking anticoagulants except low-dose aspirin)
* Increased risk for postsurgical infection (e.g., taking immunosuppressants, having a severe infection, or a having a history of serious infection)
* Known allergy to lidocaine or other anesthetics
* History of anemia
* Recent infection of target knee (within last month) requiring antibiotics
* History of bone marrow harvest or biopsy at any time
* Active malignancy or history of bone marrow malignancy

Related to previous OA management:

* Previous corticosteroid injection in the target knee within the last 3 months
* Previous viscosupplementation injection in the target knee within the last 6 months
* Previous PRP or stem cell injection in the target knee
* Previous surgery in the target knee within the last 12 months
* Previous partial or total knee replacement of the target knee
* Recent or planned surgery in the lower extremity of the target knee within 6 months

Related to other personal factors:

* Impaired cognition that impacts the ability to give informed consent
* Intense fear of needles
* Intense fear of small, enclosed spaces (i.e., claustrophobia)
* Unable to remain still for duration of MRI procedure without a sedative or anesthetic
* Likely unable to attend follow-up study visits over 6 months while enrolled in the study

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Physical Activity | Change in physical activity from baseline to 3 months.
  The investigators will use the Actigraph GT3X (Actigraph LLC, Pensacola, FL) to objectively measure physical activity. The Actigraph GT3X is a hip-worn accelerometer that measures the intensity of physical activity on a minute-by-minute basis. The Actigraph GT3X is valid and reliable in community-dwelling older adults with knee OA.

SECONDARY OUTCOMES:
Pain of Target Knee | Change in pain of target knee from baseline to 3 weeks, and change in pain of target knee from baseline to 3 months.
  The investigators will ask participants to complete the Visual Analog Scale (VAS), a single-item instrument in which the participant makes a mark on a 100 mm line to indicate their pain score in each knee from 0-100. A higher score indicates greater pain intensity of the target knee. The instrument takes <1 minute to complete.
Function of Target Knee | Change in function of target knee from baseline to 3 weeks, and change in function of target knee from baseline to 3 months.
  The investigators will ask participants to complete the Knee Injury and Osteoarthritis Outcome Score (KOOS), a 42-item instrument that assesses the following five domains: pain, symptoms (other than pain), function in activities of daily living, function in sport and recreation, and quality of life. The score is a percentage score from 0 to 100, 0 representing extreme problems of the target knee and 100 representing no problems of the target knee. The instrument takes approximately 10 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel K White, PT, ScD, MSc, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No